CLINICAL TRIAL: NCT00510770
Title: Continuous Positive Airway Pressure for Treatment of Postoperative Hypoxemia in Liver Transplant
Brief Title: CPAP in Liver Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPAP-1-LT
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Hypoxemia
Keywords: CPAP; Post-opreative; ARF; liver transplant; Post-operative hypoxemia in liver transplant
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP application

SUMMARY:
The purpose of this study is to determine the effectiveness of continuous positive airway pressure compared to standard treatment in preventing the need for intubation and mechanical ventilation in patients who develop acute hypoxemia after liver transplant.

Hypoxemia complicates the recovery of 30-50 % of patients after abdominal surgery; endotracheal intubation and mechanical ventilation may be required in 8-10 % of cases increasing morbidity and mortality and prolonging intensive care unit and hospital stay.

DETAILED DESCRIPTION:
Recovery from abdominal surgery is usually fast and uncomplicated but postoperative hypoxemia complicates 30-50 % of cases even in uneventful procedures (1). Although oxygen administration and incentive spirometry are effective in treating the vast majority of postoperative hypoxemia cases (2), respiratory failure may occur early in the postoperative course (3) requiring endotracheal intubation and mechanical ventilation in 8-10 % of patients thus increasing morbidity and mortality and prolonging intensive care unit and hospital stay (1-4). Loss of functioning alveolar units has been recognized as the underlying mechanism responsible for postoperative hypoxemia (5-7); pulmonary atelectasis after abdominal surgery is, in fact, common, it may exceed 25 % of the total lung volume and is seen several days after surgery (5-7).

Continuous positive airway pressure (CPAP) is a breathing mode where the patient spontaneously breathes through a pressurized circuit against a threshold resistor that maintains a preset positive airway pressure during both inspiration and expiration. Although several studies have demonstrated the efficacy of CPAP to reduce atelectasis and improve oxygenation in patients after abdominal surgery (8-11), no clinical trials have confirmed that the improvement of gas exchange with CPAP actually results in a reduced need for intubation and mechanical ventilation in patients who develop hypoxemia after abdominal surgery (12). We conducted a multi-center, prospective, randomized clinical trial to compare the efficacy of CPAP with standard oxygen therapy in the treatment of postoperative hypoxemia. The present study set out to examine the hypothesis that early application of CPAP may prevent intubation and mechanical ventilation in patients who develop acute hypoxemia after liver transplant.

Concealed randomization was conducted centrally through a dedicated web site using a computer-generated block randomization schedule.

Patients were randomized to be treated for six hours with oxygen through a Venturi mask at a FiO2 of 0.5 (control) or with oxygen at a FiO2 of 0.5 plus a CPAP of 7.5 cm H2O (CPAP). At the end of the 6-hour period, patients passed a one-hour screening test breathing oxygen through a Venturi mask at a FiO2of 0.3. Patients returned to the assigned treatment if the PaO2/FiO2 ratio was less than or equal to 300; treatment was interrupted if the PaO2/FiO2 ratio was higher than 300. Nasal oxygen (8-10 liter/minute) was given if the treatment was not tolerated (Figure 1).

In all centers, CPAP was generated using a flow generator with an adjustable inspiratory oxygen fraction set to deliver a flow of up to 140 liters per minute (Whisperflow, Caradyne, Ireland) and a spring-loaded expiratory pressure valve (Vital Signs Inc, Totoma NJ) and applied using a latex-free polyvinyl chloride transparent helmet (CaStar, Starmed, Italy) (15); all centers measured the inspiratory oxygen fraction using an oxygen analyzer (Oxicheck, Caradyne, Ireland) through the Venturi mask or the helmet.

All analyses were conducted on an intention-to-treat basis. Values are reported as mean and standard deviation. Continuous variables were compared with the use of the unpaired t-test or the Wilcoxon rank-sum test, depending on their distributional characteristics. Categorical variables were compared with the use of Fisher's exact test or the chi-square test, when appropriate. The Kaplan-Meier curve for intubation rate was plotted and was compared by the log-rank and Wilcoxon tests. All reported P values are two-sided.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if developed an arterial oxygen tension to inspiratory oxygen fraction ratio (PaO2/FiO2) less than or equal to 300

Exclusion Criteria:

* Age older than 80 years or younger than 18 years
* New York Heart Association functional class II III or IV
* Valvular heart disease, history of dilated cardiomyopathy, implanted cardiac pace-maker, unstable angina or myocardial infarction/cardiac surgery within the previous three months
* History of chronic obstructive pulmonary disease or asthma
* History of sleep disorders
* Preoperative infection and/or sepsis (13)
* Body mass index higher than 40
* Presence of tracheostomy, facial, neck, or chest wall abnormalities
* Requirement of emergency procedure (operation that must be performed as soon as possible and no longer than 12 hours after admission)
* Abdominal aortic aneurysm surgery
* Chemotherapy or immunosuppressive therapy within the previous three months.
* Patients were also excluded if before randomization they showed:

  * Arterial pH lower than 7.30 with an arterial carbon dioxide tension higher than 50 mmHg
  * Arterial oxygen saturation lower than 80 % with the maximal fraction of inspiratory oxygen; clinical signs of acute myocardial infarction
  * Systolic arterial pressure lower than 90 mmHg under optimal fluid therapy
  * Presence of criteria for acute respiratory distress syndrome (14)
  * Hemoglobin concentration lower than 7 g/dl, serum albumin lower than 3 g/dl
  * Creatinine level higher than 3.5 g/dl
  * Glasgow Coma Scale lower than 12.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-12

PRIMARY OUTCOMES:
Intubation, need of mechanical ventilation

SECONDARY OUTCOMES:
Wound infection, ICU Los , Hospital Los

CONTACTS AND LOCATIONS:
Overall Officials: Squadrone SV Vincenzo, MD, Principal Investigator
Locations (1):
- Università degli Studi Torino, Turin, Piedmont, Italy